CLINICAL TRIAL: NCT00722735
Title: A Double-Blind, Double-Dummy, Prospective, Randomized Multiple-Site Study of Oral Finafloxacin 300 mg b.i.d. Versus Oral Ciprofloxacin 250 mg b.i.d. in Patients With Lower Uncomplicated UTI (uUTI) With a Treatment Duration of 3 Days
Brief Title: Finafloxacin 300 mg Twice a Day (b.i.d.) Versus Ciprofloxacin 250 mg Twice a Day (b.i.d) in Patients With Lower Uncomplicated UTI (uUTI)
Acronym: FLUT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MerLion Pharmaceuticals GmbH (Industry)
Responsible Party: Jasper Hein, MD, Prinzipal Investigator, Practicing Physician
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FINA-003
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2008-10

CONDITIONS: Urinary Tract Infections
Keywords: uncomplicated Urinary Tract Infection in Women; Antibacterial Chemotherapy; Proof-of-Concept
MeSH Terms: conditions — Urinary Tract Infections | interventions — finafloxacin; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Group I: Finafloxacin tablets + Ciprofloxacin placebo capsule
  Interventions: Drug: Finafloxacin
- 2 (Active Comparator): Group II: Ciprofloxacin capsule + Finafloxacin placebo tablets
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Finafloxacin — Finafloxacin tablets, 300 mg b.i.d., oral administration; Ciprofloxacin placebo capsule, 1 capsule b.i.d.,oral administration; duration: 3 days
  Arms: 1
Drug: Ciprofloxacin — Finafloxacin placebo, 6 tablets b.i.d., oral administration; Ciprofloxacin capsule, 250 mg b.i.d., oral administration; duration: 3 days
  Arms: 2

SUMMARY:
To compare the bacteriological eradication rates of Finafloxacin and Ciprofloxacin in female patients with uUTI.

DETAILED DESCRIPTION:
Patients with clinical signs and symptoms of uUTI who have a high probability of the required number of bacteria in their urine, measured by positive test for nitrite and /or leucocyte esterase by means of a dipstick will be enrolled in this study. Only these patients with bacterial count equal or more than 10e5 cfu/mL will be included in the efficacy analysis. At Baseline, patients will be randomly assigned (2:1) to receive Finafloxacin 300 mg or Ciprofloxacin 250 mg, following a double-dummy design, ie Group 1 will receive Finafloxacin tablets + Ciprofloxacin placebo capsule while Group II will receive Ciprofloxacin capsule + Finafloxacin placebo tablets. The treatment will last in total 3 days. The microbiological results will be compared with the baseline microbiology. If the concentration of initial pathogen in the urine is equal or more than 10e3 cfu/mL in the post-therapy culture compared with the baseline , this will define a bacteriological eradication. Microbiological assessment will be performed as well. Evaluation of the bacteria reinfection or relapse will be performed, based on the microbiology results. The status of clinical improvement and cure will be considered additionally.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients between 18 and 55 years with uUTI.
2. Two of the following sign and symptoms of uUTI: dysuria, frequency, urgency, miction pain, suprapubic pain, gross hematuria, turbid urine or malodorous urine.
3. Able to supply a mid-stream, clean catch urine sample for microbiological analysis.
4. The result of the dipstick should indicate a high probability of the required number of bacteria.
5. Be able to communicate with the study personnel.
6. Has given written consent to participate in the study.

Exclusion Criteria:

1. Female patients having signs and symptoms of upper urinary tract infection (e.g. fever, flank pain) indicating complicated UTI.
2. Male patients
3. History or evidence of other functional or anatomical abnormalities of the urinary tract (e.g. acute pyelonephritis), diabetes mellitus and immunosuppression.
4. Recurrent cystitis with more than 3 episodes in the past 12 months.
5. Clinical symptoms for more than 7 days before Baseline.
6. Psychiatric, neurological or behavior disorders.
7. Clinically significant serious unstable physical illness.
8. Known uncontrolled condition of hypertension or symptomatic hypotension, known ischemic heart disease or history of myocardial infarction (within 12 months prior study enrolment), coronary artery bypass surgery or percutaneous transluminal coronary angioplasty.
9. Existence of any surgical or medical condition which might interfere with the distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract.
10. Antibiotic intake 2 weeks before study enrolment.
11. Failed UTI therapy within 2 months before study inclusion.
12. Expectancy of concomitant administration of antibiotics, sucralfate or divalent and trivalent cations such as iron or antacids containing magnesium, aluminium or calcium intake during the course of the study.
13. Clinically abnormal vital signs, ECG findings and safety laboratory results at Baseline.
14. Known hypersensitivity or contraindication to the use of fluoroquinolones.
15. History of tendon lesions or ruptures during quinolone treatment.
16. Any malignant disease or a history of malignant neoplasm other than carcinoma in situ of the cervix or basal cell carcinoma of the skin, within the last 5 years before Baseline.
17. Current diagnosis or history of substance abuse.
18. Exposure to any of the investigational drugs 30 days prior to Baseline.
19. Pregnant or nursing woman, or woman of childbearing potential who is not using an effective contraceptive method during the study, e.g. oral (stable doses for at least 3 months prior to Baseline) or injectable (stable doses for at least 2 months prior to Baseline) contraceptives, intrauterine devices (for at least 2 months prior Baseline), double-barrier method, contraceptive patch, female sterilization or condoms.
20. The patient, planned to be enrolled is an employee of any involved study investigator or any involved institution including the study sponsor.
21. Inability or lacking motivation to participate in the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Bacteriological eradication of the initial pathogen. | 4-6 days

SECONDARY OUTCOMES:
Clinical cure: Absence of signs or symptoms of uUTI. | 10-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Hein, MD, Principal Investigator
Locations (2):
- Medical practice, Dr. J. Hein (Principal Study Investigator), Marburg, Germany
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Vente A, Bentley C, Luckermann M, Tambyah P, Dalhoff A. Early Clinical Assessment of the Antimicrobial Activity of Finafloxacin Compared to Ciprofloxacin in Subsets of Microbiologically Characterized Isolates. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e02325-17. doi: 10.1128/AAC.02325-17. Print 2018 Apr. PMID 29339393